CLINICAL TRIAL: NCT03589781
Title: Investigating the Effects of Mikei® Red Reishi Essence EX on the Immune System of Prostate Cancer Patients and Patients With Non-cancerous Conditions of the Prostate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid 19 Pandemic - Unable to enroll patients
Sponsor: Nikkei (Canada) Marketing Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RM5160
Record Dates: First submitted 2018-05-16; First posted 2018-07-18 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mikei Red Reishi Essence EX (Experimental): There are two groups (50 participants total) in this clinical study, one group (35 participants) will be given Mikei® Red Reishi Essence EX product (Product Group).
  Interventions: Dietary Supplement: Mikei Red Reishi Essence EX
- Placebo (Placebo Comparator): Another group (15 participants) will be given the placebo (Placebo Group). Placebo is a pill that looks like a drug but has no drug or other active ingredients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mikei Red Reishi Essence EX — Dosage is 490 mg per capsule, 3 capsules twice a day with food or water. Total of 6 capsules per day.
  Other Names: Ganoderma lucidum (fruiting body) extract; lingzhi
  Arms: Mikei Red Reishi Essence EX
Dietary Supplement: Placebo — Matching placebo. Consume 3 capsules twice a day with food or water. Total of 6 capsules per day.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effects of Mikei® Red Reishi Essence EX extract powder on the immune function of prostate cancer patients and patients with non-cancerous conditions of the prostate.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of Mikei® Red Reishi Essence EX, a natural supplementary dietary product, on the immune function of prostate cancer patients and patients with non-cancerous conditions of the prostate. According to limited published scientific research and clinical studies, Reishi mushroom extract may support the body's immune function. According to cancer immunology research, at early stage of tumor development, the immune system can mount defensive actions to eliminate or inhibit tumor growth. This study is to examine the specific effect of Mikei® Red Reishi Essence EX on the immune function of prostate cancer patients and patients with non-cancerous conditions of the prostate.

ELIGIBILITY:
Inclusion Criteria:

1. Male age between 50-85
2. Diagnosed with prostate cancer or high-grade PIN within the last 24 months through the most recent biopsy; or patients who have a total PSA level above 4.0 but have not been diagnosed with prostate cancer yet
3. Has not received any prostate cancer therapy including surgery, chemotherapy, hormone therapy, or radiation therapy
4. Clinical Gleason score of the tumor is ≤6 for patients ≤70 years or ≤7 for >70 years; (non-applicable for non-cancer patients with elevated PSA or high-grade PIN)
5. The clinical stage of the cancer is T1c or below (non-applicable for non-cancer patients with elevated PSA or high-grade PIN)
6. The patients have been recommended for and placed under active surveillance without immediate treatment
7. Able to provide written informed consent

Exclusion Criteria:

1. Patients taking mushroom (including reishi) or other herbal products/natural supplements
2. Patients with a known allergy to mushrooms
3. Prisoners
4. Patients who receive treatment with 5-alpha reductase inhibitors (finasteride [Propecia®, Proscar®,], or dutasteride [Avodart®) within 28 days prior to randomization are not eligible. The use of these drugs is not allowed during the patients' study participation.
5. Patients with a history of non-cutaneous malignancy in the previous 5 years are not eligible.
6. Patients taking warfarin, heparin, Aspirin >81mg/day, or other prescribed blood thinners: Reishi may increase the risk of bleeding.
7. Patients with platelets levels below 139 X 103/ul or history of bleeding disorders
8. Patients undergoing chemotherapy: Reishi may make some chemotherapy drugs less effective.
9. Patients with any known immune disorder, including but not limited to HIV or other primary or secondary immune deficiency diseases, autoimmune diseases, history of or being considered for organ transplants, etc.
10. Patients taking immunosuppressants (Corticosteroids, Calcineurin inhibitors, mTOR inhibitors, IMDH inhibitors, Biologics, Monoclonal antibodies): Reishi can stimulate immune responses.
11. Patients taking cytochrome P450 2E1, 1A2, and 3A sensitive substrate drugs: Reishi may increase the risk of side effects of these drugs.
12. Patient has total bilirubin >1.5 MG/DL, alanine aminotransferase (ALT) >51 U/L or aspartate aminotransferase (AST) >46 U/L.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-05 (Estimated); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in the immune function of the prostate cancer patients and patients with non-cancerous prostate conditions by taking reishi extract product. The immune function will be analyzed using D2Dx test by measuring the relative IgG level in the blood. | 6 months
  D2Dx test is a two-step blood test that can measure the amount of IgG antibody adsorbed to a gold nanoparticle. Using a goat anti-human IgG antibody, the relative amount of IgG against autoantibodies is detected.

SECONDARY OUTCOMES:
Correlation between the immune function as expressed in the IgG level in the blood and the disease status (determined by PSA, DRE changes, and Gleason score) of prostate cancer patients. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Inoel Rivera, MD, Principal Investigator — Orlando Health Medical Group Urology; Qun Huo, Ph.D., Principal Investigator — University of Central Florida
Locations (1):
- Orlando Health Medical Group Urology, Orlando, Florida, United States